CLINICAL TRIAL: NCT05863767
Title: Effect of Baduanjin Sequential Therapy on Physical Functioning and Quality of Life Among Post CABG Patients.
Brief Title: Effects of Baduanjin Sequential Therapy on Post CABG Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01387 Iqra Ayub
Record Dates: First submitted 2023-04-12; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Post-cardiac Surgery
Keywords: Baduanjin sequential therapy; CABG; Physical functioning; Quality of life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Baduanjin sequential therapy consists of Six different movements including the preparatory phase. The session will account for 30 minutes twice a day for four weeks.
  Interventions: Other: Baduanjin sequential therapy
- Control group (Placebo Comparator): Control intervention: AROM, Breathing exercises, and stretches 5 repetitions three times a day.
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Baduanjin sequential therapy — Baduanjin sequential therapy consists of eight different movements including the preparatory phase till final movement (gathering the energy). The session will account for 30 minutes twice a day for four weeks.
  Arms: Interventional Group
Other: Conventional Therapy — Neck stretches Arm circles Triceps stretch Calf stretch Forward step up Strengthening exercises Every exercise 5 repetitions three times a day
  Arms: Control group

SUMMARY:
To determine the effects of Baduanjin sequential therapy (BST) on physical functioning and quality of life among post-CABG patients. Many studies have focused on the effects of standing Baduanjin on chronic diseases and it's an evidence-based therapy.

DETAILED DESCRIPTION:
There exists limited data from large-scale randomized trials that have addressed the effect of Baduanjin exercise on the quality of life and cardiac function in the patient with CABG. Therefore, this study aims to determine the effects of Baduanjin sequential therapy (BST) on physical functioning and quality of life among post-CABG patients.

ELIGIBILITY:
Inclusion Criteria:

* Vitally Open heart surgery patients Discharged from the hospital and enrolled as outpatient Able to perform 6MWT

Exclusion Criteria:

* Prolonged intubation Unstable vitals Patient needs maximum assistance for mobility Decline consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | 4 weeks
  Changes from baseline to 4 weeks, measured through 6 min walk test (6 MWT) used to measure Functional capacity. It is a submaximal exercise test that can aid in assessing the functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters that an individual covers in 6 min without any support.
Functional performance | 4 weeks
  Changes from baseline to 4 weeks, measured through Short physical performance battery. It is a commonly used tool in clinical setting for measuring the physical performance of patients. It is divided into three subtests: balance, a short walk at normal pace and lastly standing up from a chair five times repeatedly. These subsets exemplify core tasks being important for independent living. Scoring of each test range from s 0 (worst performance) to 4 (best performance). The sum total for the entire battery is between 0 to 12 which is the sum of all 3 tests. The cutoff point is 10 or lower for mobility impairment. Low scores on shows health consequences related with disability in Activities of Daily Living.
Health related Quality of Life (QOL) | 4 weeks
  Changes from baseline to 4 weeks, measured through Short Form 36 Health Survey Questionnaire (SF-36) that is used to indicate the health status of a particular population. This tool consists of eight domains comprising functional capability, role physical functioning, role emotional functioning, psychological state, liveliness, social affairs, bodily pain, and overall health. Responses are marked on a Likert scale comprising of 5 points and then converted on a scale of 100. Attaining scores more than 50 indicated a better state of health and the lower score the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Peshawar Institute of cardiology, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mao S, Zhang X, Chen M, Wang C, Chen Q, Guo L, Zhang M, Hinek A. Beneficial Effects of Baduanjin Exercise on Left Ventricular Remodelling in Patients after Acute Myocardial Infarction: an Exploratory Clinical Trial and Proteomic Analysis. Cardiovasc Drugs Ther. 2021 Feb;35(1):21-32. doi: 10.1007/s10557-020-07047-0. Epub 2020 Aug 6. PMID 32761487
- [Background] Chen MG, Liang X, Kong L, Wang J, Wang F, Hu X, He J, Zeng RX, Mao S, Guo L, Zhang MZ, Zhang X. Effect of Baduanjin Sequential Therapy on the Quality of Life and Cardiac Function in Patients with AMI After PCI: A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2020 Jul 4;2020:8171549. doi: 10.1155/2020/8171549. eCollection 2020. PMID 32714423
- [Background] Chen DM, Yu WC, Hung HF, Tsai JC, Wu HY, Chiou AF. The effects of Baduanjin exercise on fatigue and quality of life in patients with heart failure: A randomized controlled trial. Eur J Cardiovasc Nurs. 2018 Jun;17(5):456-466. doi: 10.1177/1474515117744770. Epub 2017 Nov 30. PMID 29189045